CLINICAL TRIAL: NCT02639065
Title: A Phase II Study Evaluating Safety and Efficacy of Durvalumab (MEDI4736) Following Multi-modality Therapy in Esophageal Cancer: Big Ten Cancer Research Consortium BTCRC-ESO14-012
Brief Title: A Study of Durvalumab (MEDI4736) in Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shadia Jalal, MD (Other)
Collaborators: MedImmune LLC (Industry); AstraZeneca (Industry); Big Ten Cancer Research Consortium (Other)
Responsible Party: Sponsor-Investigator, Shadia Jalal, MD, Sponsor-Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-ESO14-012
Record Dates: First submitted 2015-12-21; First posted 2015-12-24 (Estimated); Results first posted 2022-06-01 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Esophageal Cancer
Keywords: Durvalumab; MEDI4736; PD-L1 inhibitor
MeSH Terms: conditions — Esophageal Neoplasms | interventions — durvalumab

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigational Treatment (Experimental): Durvalumab 1500 mg IV every 4 weeks (1 cycle) for a maximum 13 doses (12 months), or until unacceptable toxicities or disease recurrence.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — 1500 mg IV every 4 weeks (1 cycle) for a maximum 13 doses (12 months), or until unacceptable toxicities or disease recurrence.
  Other Names: MEDI4736

SUMMARY:
This is a phase II, open-label, single arm, single-stage study. A total of 23 evaluable patients will be enrolled. If total number of patients free of disease relapse at 1 year is less than or equal to 15, the drug would not be considered for further study in this setting. After six patients are treated with at least one dose of study drug, they will be observed for a minimum of 60 days. During the 60-day observation period, further accrual will be halted to evaluate "unacceptable toxicities warranting early closure of the trial" defined as:

* Any definitive durvalumab-related death. A durvalumab-related death will be continuously monitored throughout the trial and the trial will be suspended for re-evaluation whenever such an event is confirmed.
* Any unexpected and previously unreported grade 4 toxicities definitely related to durvalumab.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center trial.

INVESTIGATIONAL TREATMENT:

Subjects will receive durvalumab 1500 mg IV every 4 weeks (1 cycle) for a maximum 13 doses (12 months), or until unacceptable toxicities or disease recurrence.

The following baseline labs must be completed within 28 days prior to registration for protocol therapy:

Hematopoietic:

* White blood cell count (WBC) > 3 K/mm^3
* Hemoglobin (Hgb) > 9 g/dL. Transfusion is allowed, if needed, since patients are post esophagectomy.
* Platelets > 100 K/mm^3
* Absolute neutrophil count (ANC) ≥ 1.5 K/mm^3

Renal:

* Calculated creatinine clearance of >/= 40 cc/min using the Cockcroft-Gault formula or by 24-hour urine collection.

Hepatic:

* Bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST, SGOT) </= 2.5 x ULN
* Alanine aminotransferase (ALT, SGPT) </= 2.5 x ULN

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of protected health information obtained from the subject prior to performing any protocol-related procedures, including screening evaluations. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0-1 within 28 days prior to registration for protocol therapy.
* Females of childbearing potential and males must be willing to use two effective methods of contraception (see the protocol) from the time consent is signed until 3 months after treatment discontinuation.
* Females of childbearing potential must have a negative serum pregnancy test within 14 days prior to registration for protocol therapy. NOTE: Female subjects are considered of child bearing potential unless they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are ≥60 years old and naturally postmenopausal for at least 12 consecutive months. See the protocol.
* Histological evidence of persistent residual esophageal adenocarcinoma including gastroesophageal junction adenocarcinoma following definitive concurrent chemoradiotherapy (carboplatin and paclitaxel or cisplatin and 5-FU) in the surgical sample (esophagus or lymph node or both) obtained at the time of esophagectomy. NOTE: Persistent residual disease is defined as follows (modified from College of American Pathologists Guidelines):

  * No residual tumor (Grade 0, complete response, 0% tumor). This group will not be included in this study.
  * Marked response (Grade 1, 0-<10% residual tumor)
  * Moderate response (Grade 2, 10-50% residual tumor)
  * No definite response (Grade 3, >50% residual tumor)
* Minimum of 1 month and maximum of 3 months from surgical resection with no evidence of disease progression at the time of enrollment.
* Must have adequately recovered from surgery as judged by the treating investigator.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Prior therapy with a PD-1, PD-L1, or CTLA-4 inhibitor or cancer-specific vaccine therapy.
* Evidence of active autoimmune disease requiring systemic treatment within preceding 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Exceptions to this rule include vitiligo, resolved childhood asthma/atopy, requirement of intermittent bronchodilators or local steroid injections, hypothyroidism stable on hormone replacement, psoriasis not requiring systemic treatment (within the past 2 years), Graves's disease and Sjogren's syndrome.
* Prior malignancy is not allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, Gleason score ≤ 7 prostate cancers, or other cancer for which the subject has been disease-free for at least 3 years.
* Active or prior documented inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis).
* Presence of interstitial lung disease or history of pneumonitis requiring treatment with corticosteroids.
* Patients with diagnosis of primary immunodeficiency.
* Patients receiving chronic systemic corticosteroid therapy or other immunosuppressive therapy within 28 days prior to registration for protocol therapy. Exceptions include intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
* History of allogeneic organ or stem cell transplant.
* Receipt of live attenuated vaccine within 30 days prior to registration for protocol therapy.
* Mean QT interval corrected for heart rate (QTc) > 470 msec calculated from 3 ECGs by Bazett's Correction.
* Ventricular arrhythmias requiring medication(s).
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, or active bleeding diatheses.
* History of psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
* Known HIV infection or chronic hepatitis B or C.
* Known history of previous clinical diagnosis of tuberculosis.
* Clinically significant infections as judged by the treating investigator. Clinically significant is defined as an active infection requiring IV antibiotics.
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued. In addition, breast milk cannot be stored for future use while the mother is being treated on study.
* Treatment with any investigational agent within 28 days prior to registration for protocol therapy.
* History of hypersensitivity to durvalumab or any excipient.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
* Previous enrollment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2021-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shadia Jalal, M.D., Study Chair — Big Ten Cancer Research Consortium
Locations (3):
- United States (3):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Unversity of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Michigan Health System, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mamdani H, Schneider B, Perkins SM, Burney HN, Kasi PM, Abushahin LI, Birdas T, Kesler K, Watkins TM, Badve SS, Radovich M, Jalal SI. A Phase II Trial of Adjuvant Durvalumab Following Trimodality Therapy for Locally Advanced Esophageal and Gastroesophageal Junction Adenocarcinoma: A Big Ten Cancer Research Consortium Study. Front Oncol. 2021 Sep 17;11:736620. doi: 10.3389/fonc.2021.736620. eCollection 2021. PMID 34604072
- See also: Big Ten Cancer Research Consortium Website — http://www.bigtencrc.org

RESULTS

PARTICIPANT FLOW:
Period: Study Treatment
Arm/Group | Investigational Treatment
Started | 39
Completed | 16
Not Completed | 23
Not completed — Disease Progression | 13
Not completed — Adverse Event | 9
Not completed — Withdrawal by Subject | 1
Period: Follow up
Arm/Group | Investigational Treatment
Started | 39
Completed | 30
Not Completed | 9
Not completed — Subject refused to follow up | 1
Not completed — Symptomatic Deterioration | 2
Not completed — Death | 2
Not completed — Study Terminated | 1
Not completed — Disease Progression | 3

BASELINE CHARACTERISTICS:
Population: This population includes all subjects who were enrolled and found eligible and evaluable for this trial.
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 37
Age, Customized [Median (Full Range); unit: years] | 61 [43 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 37
  Race: Unknown | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 1
  Ethnicity: Non-Hispanic | 35
  Ethnicity: Unknown | 1
Site [Count of Participants; unit: Participants]
  Indiana University | 25
  University of Iowa | 5
  University of Michigan | 7
Site of Disease [Count of Participants; unit: Participants]
  Gastroesophageal Junction | 18
  Distal Esophagus | 19
Chemotherapy Regimen [Count of Participants; unit: Participants]
  Cisplatin + 5FU | 6
  Carboplatin + paclitaxel | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With One-Year Relapse Free Survival (RFS) With Post-Operative Durvalumab
Description: Relapse free survival is defined as time from the date of surgery until the criteria for disease relapse is met, per Response Evaluation Criteria In Solid Tumors (RECIST 1.1), or death occurs.
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started The percentage of subjects who attained relapse free survival for 1 year and 95 % confidence interval has been reported here.
Time Frame: From the date of surgery until disease relapse or death up to a maximum of 40 months.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 37
percentage of subjects | 73 [56 to 84]

2. Secondary Outcome: Number of Patients With Adverse Events as a Measure of Safety and Tolerability
Description: One of the secondary objective in this study is to assess toxicity and tolerability of durvalumab following trimodality therapy in patients with esophageal cancer. Adverse events were recorded from the time of consent for at least 90 days after treatment discontinuation, per Common Terminology Criteria for Adverse Events (CTCAE) v4. Events were assessed at every visit at an interval of 4 weeks.
  Adverse Event severity grades can be described as follows :
  * Grade 1 indicates a mild event
  * Grade 2 indicates a moderate event
  * Grade 3 indicates a severe event
  * Grade 4 indicates a potentially life-threatening event
  * Grade 5 indicates death
Time Frame: From the time of consent until 90 days after last dose of durvalumab up to a maximum of 15 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 37
Participants
  Patient had at least one adverse event of any grade | 37
  Patient had at least one grade 3 or greater adverse event | 22
  Patient had at least one grade 3 or greater treatment related adverse event | 10
  Patient having serious adverse event | 9

3. Post Hoc Outcome: Median Relapse Free Survival.
Description: Relapse free survival is defined as time from the date of surgery until the criteria for disease relapse is met, per Response Evaluation Criteria In Solid Tumors (RECIST 1.1), or death occurs.
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started Here Median Relapse Free Survival time in months has been reported.
Time Frame: From the date of surgery until disease relapse or death up to a maximum of 40 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 37
months | 21.0 [14.0 to 40.4]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of consent until 90 days after last dose of durvalumab up to a maximum of 15 months.
Description: Adverse events were recorded from the time of consent for at least 90 days after treatment discontinuation, per Common Terminology Criteria for Adverse Events (CTCAE) v4. Events were assessed at every visit at an interval of 4 weeks.
Arm/Group | Investigational Treatment
All-Cause Mortality (participants affected / at risk) | 2/37
Serious Adverse Events (participants affected / at risk) | 9/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Treatment (N=37)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
ENCEPHALOPATHY (Nervous system disorders) | 1 (2)
HEMATURIA (Renal and urinary disorders) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
LUNG INFECTION (Infections and infestations) | 2 (3)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PSYCHIATRIC DISORDERS - OTHER, SPECIFY (Psychiatric disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Treatment (N=37)
ABDOMINAL INFECTION (Infections and infestations) | 1 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (7)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5 (10)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 (4)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
ANEMIA (Blood and lymphatic system disorders) | 7 (11)
ANOREXIA (Metabolism and nutrition disorders) | 8 (9)
ANXIETY (Psychiatric disorders) | 4 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 9 (16)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 6 (16)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (8)
BLOOD AND LYMPHATIC SYSTEM DISORDERS (Blood and lymphatic system disorders) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 3 (8)
BURN (Injury, poisoning and procedural complications) | 1 (1)
CARDIAC DISORDERS (Cardiac disorders) | 1 (1)
CHEST PAIN - CARDIAC (Cardiac disorders) | 1 (1)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CHILLS (General disorders) | 2 (5)
CHOLESTEROL HIGH (Investigations) | 1 (1)
COLITIS (Gastrointestinal disorders) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 5 (5)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (7)
CREATININE INCREASED (Investigations) | 3 (6)
DENTAL CARIES (Gastrointestinal disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 16 (34)
DIZZINESS (Nervous system disorders) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 3 (3)
DYSPEPSIA (Gastrointestinal disorders) | 1 (2)
DYSPHAGIA (Gastrointestinal disorders) | 9 (10)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 4 (4)
EAR PAIN (Ear and labyrinth disorders) | 1 (1)
ELECTROCARDIOGRAM QT CORRECTED INTERVAL PROLONGED (Investigations) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 2 (4)
FATIGUE (General disorders) | 13 (21)
FECAL INCONTINENCE (Gastrointestinal disorders) | 1 (1)
FEVER (General disorders) | 2 (2)
FLATULENCE (Gastrointestinal disorders) | 1 (1)
FLU LIKE SYMPTOMS (General disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 (3)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 1 (2)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (4)
HEADACHE (Nervous system disorders) | 4 (4)
HEMATURIA (Renal and urinary disorders) | 3 (5)
HEMORRHOIDS (Gastrointestinal disorders) | 2 (2)
HEPATOBILIARY DISORDERS (Hepatobiliary disorders) | 1 (1)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HOT FLASHES (Vascular disorders) | 1 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 2 (6)
HYPERPARATHYROIDISM (Endocrine disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 6 (6)
HYPERTHYROIDISM (Endocrine disorders) | 3 (3)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 2 (3)
HYPOKALEMIA (Metabolism and nutrition disorders) | 4 (7)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1)
INFUSION SITE EXTRAVASATION (General disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 4 (4)
INVESTIGATIONS (Investigations) | 3 (4)
LOCALIZED EDEMA (General disorders) | 1 (1)
LUNG INFECTION (Infections and infestations) | 5 (6)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1)
METABOLISM AND NUTRITION DISORDERS (Metabolism and nutrition disorders) | 1 (1)
MUSCLE WEAKNESS TRUNK (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 8 (12)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 12 (22)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (2)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 2 (3)
NEURALGIA (Nervous system disorders) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2)
PAIN (General disorders) | 3 (5)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (2)
PARESTHESIA (Nervous system disorders) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 (3)
PLATELET COUNT DECREASED (Investigations) | 2 (2)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PROTEINURIA (Renal and urinary disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 6 (7)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 (2)
RASH PUSTULAR (Infections and infestations) | 1 (1)
RENAL CALCULI (Renal and urinary disorders) | 1 (3)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1)
SERUM AMYLASE INCREASED (Investigations) | 2 (7)
SICK SINUS SYNDROME (Cardiac disorders) | 1 (1)
SINUSITIS (Infections and infestations) | 2 (3)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN INFECTION (Infections and infestations) | 1 (1)
STOMACH PAIN (Gastrointestinal disorders) | 2 (3)
SURGICAL AND MEDICAL PROCEDURES (Surgical and medical procedures) | 3 (3)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3)
URINE DISCOLORATION (Renal and urinary disorders) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 7 (11)
WEIGHT GAIN (Investigations) | 3 (4)
WEIGHT LOSS (Investigations) | 8 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT02639065/Prot_SAP_000.pdf